CLINICAL TRIAL: NCT02102139
Title: A Single Preoperative Injection of Dexmedetomidine Attenuates Haemodynamic Responses to Hydrodissection in Patients Undergoing Robotic Thyroidectomy: a Prospective Randomised Double-blinded Study
Brief Title: Preop Dexmedetomidine Attenuates Haemodynamic Responses to Hydrodissection
Acronym: DXM_Hydro
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Hee-Pyoung Park, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Supportive Care
Other Study IDs: DXM_Hydrodissection
Record Dates: First submitted 2014-03-26; First posted 2014-04-02 (Estimated); Last update posted 2014-04-02 (Estimated); Status verified 2014-03

CONDITIONS: Robotic Thyroidectomy
MeSH Terms: interventions — Propofol; Sodium Chloride

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- DXM + Propofol (Experimental): DXM (1 µg kg -1) was loaded intravenously for 10 min before anaesthesia induction.During DXM loading, the depth of anaesthesia was monitored using a bispectral index (BIS) monitor. Electrocardiogram, heart rate, pulse oximetry, and non-invasive arterial blood pressure were monitored at 2-min intervals.
  Anaesthesia was induced with propofol 3.5 μg mL 1 and remifentanil 5 ng mL 1 at an effect site concentration using a target-controlled infusion (TCI) device. Anaesthesia was maintained with propofol and remifentanil continuous infusions.
  During surgery except the study period, propofol and remifentanil doses were adjusted to maintain BIS value of 40-60 and systolic blood pressure (SBP) within ±20% from baseline respectively.
  Interventions: Drug: DXM + Propofol
- Saline + Propofol (Placebo Comparator): Saline (1 µg kg -1) was loaded intravenously for 10 min before anaesthesia induction.During saline loading, the depth of anaesthesia was monitored using a bispectral index (BIS) monitor. Electrocardiogram, heart rate, pulse oximetry, and non-invasive arterial blood pressure were monitored at 2-min intervals.
  Anaesthesia was induced with propofol 3.5 μg mL 1 and remifentanil 5 ng mL 1 at an effect site concentration using a target-controlled infusion (TCI) device. Anaesthesia was maintained with propofol and remifentanil continuous infusions.
  During surgery except the study period, propofol and remifentanil doses were adjusted to maintain BIS value of 40-60 and systolic blood pressure (SBP) within ±20% from baseline respectively.
  Interventions: Drug: Saline + Propofol

INTERVENTIONS:
Drug: DXM + Propofol — After induction as mentioned at 'arm description', the effect-site propofol concentration was fixed at 5.0 μg mL-1 at the time of diluted epinephrine injection and was unchanged during the entire hydrodissection period in all patients.
  The first patients received effect-site concentrations of remifentanil of 4 ng mL -1, respectively. The EC50 of remifentanil for stable hydrodissection was determined by a modification of Dixon's up-and-down method.If the response was "success (SBP during the entire hydrodissection period being ±20% from baseline)," the next target concentration of remifentanil was decreased by a step of 0.5 ng mL -1. If the response was "fail(SBP > ±20% from baseline)," the target concentration was increased by 0.5 ng mL-1.
  Arms: DXM + Propofol
Drug: Saline + Propofol — All procedure would be same in DXM+Propofol group except saline loading rather than DXM loading before induction.
  Arms: Saline + Propofol

SUMMARY:
Percutaneous tunnelling (hydrodissection) in the neck and anterior chest in patients undergoing robotic thyroidectomy leads to significant haemodynamic responses such as increases in blood pressure and heart rate. The investigators evaluated whether a single preoperative dexmedetomidine injection attenuated the haemodynamic responses to hydrodissection by reducing the half-maximal effective concentration (EC50) of remifentanil needed to maintain haemodynamic stability during hydrodissection.

DETAILED DESCRIPTION:
Dexmedetomidine (DXM) is a recently released and approved alpha 2 agonist with a relatively high ratio of α2/α1-activity and an almost fourfold shorter half-life than clonidine.It's sympatholytic, sedative, and analgesic properties makes DXM a useful anaesthetic adjuvant for general anaesthesia. While there are some reports of the beneficial effects of DXM on anaesthetic requirements and haemodynamic responses to endotracheal intubation, the effect of a single preoperative injection of DXM in terms of attenuating haemodymanic responses to surgical stimulation in robot-assisted thyroidectomy is unknown.

When a robotic thyroidectomy using the bilateral axillary breast approach (BABA) technique is performed, subcutaneous tunnelling in the neck and anterior chest, which is defined as hydrodissection, is mandatory. Unfortunately, the procedure leads to significant haemodynamic responses, such as increases in blood pressure and heart rate.

We hypothesised that preoperative DXM administration would attenuate the haemodynamic responses to hydrodissection. This study was designed to evaluate the effects of a single preoperative administration of DXM on haemodynamic responses to hydrodissection in robotic thyroidectomy by comparing the half-maximal effective concentration (EC50) of remifentanil needed to maintain haemodynamic stability during hydrodissection between DXM and control groups. We also investigated the effects of preoperative DXM administration on total doses of remifentanil and propofol administered intraoperatively.

ELIGIBILITY:
Inclusion Criteria:

* ASA physical status I-II patientsscheduled for general anaesthesia for robotic thyroidectomy

Exclusion Criteria:

* Patients with an allergy to α2-adrenergic agonists or propofol
* Patients with current antihypertensive medication
* Patients with heart block > 1 degree
* Patients with severe cardiorespiratory dysfunction
* Patients with history of alcohol or drug abuse
* Patients who had received an opioid analgesic medication within the previous 24-h period before the operation

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2012-05; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Remifentanil EC50 during hydrodissection | at the time point of hydrodissection intraopeartively
  Compare remifentanil EC50 for maintaining haemodynamic stability during hydrodissection between 2 groups.
  The EC50 of remifentanil for maintaining haemodynamic stability was determined by a modification of Dixon's up-and-down method.If the response was "success (SBP during the entire hydrodissection period being ±20% from baseline)," the next target concentration of remifentanil was decreased by a step of 0.5 ng mL -1. If the response was "fail(SBP > ±20% from baseline)," the target concentration was increased by 0.5 ng mL-1.

SECONDARY OUTCOMES:
Total doses of remifentanil & propofol administration | Intraoperatively
  Compare total doses of remifentanil and propofol administered intraoperatively between 2 groups.

CONTACTS AND LOCATIONS:
Overall Officials: Hee Pyung Park, MD PhD, Study Director — Professor; Young Jin Lim, Md PhD, Principal Investigator — Professor
Locations (1):
- Seoul National University of Hospital, Seoul, South Korea